CLINICAL TRIAL: NCT03804658
Title: The Effects of Glucose Monitor on Patients With Diabetes
Brief Title: The Factors Affecting the Achievement of Glucose Monitor in the Patients on Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CG18308A
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Glucose Variability; Cognitive Decline
Keywords: Brain-derived neurotrophic factor; Vascular cell adhesion molecule 1; Renalase; Orexin; Continue glucose monitor
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Serum, Plasma and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continue glucose monitor system — The cardiovascular risks and data from continue glucose monitor system

SUMMARY:
To assess the effect of glucose monitors on glucose control and cardiovascular risks.

DETAILED DESCRIPTION:
The investigators will enroll patients with diabetes. The answered questionnaire and blood samples will be collected at baseline. After change the methods or frequency of glucose monitor, the blood samples will be collected again. The investigators will analyze the factors which may affect the glucose control after changes in methods of glucose monitor.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diabetes

Exclusion Criteria:

* Incooperative patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diabetes both in outpatient and inpatient
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucose variability | 3 months
  Data from continue glucose monitor system

SECONDARY OUTCOMES:
brain-derived neurotrophic factor | 3 months
  Biomarker of cognition
Orexin | 3 months
  Biomarker of cognition
Renalase | 3 months
  Biomarker of cognition
Vascular endothelial cell adhesion molecule 1 | 3 months
  Biomarker for inflammation
Health Literacy | 3 months
  Questionnaire of health

CONTACTS AND LOCATIONS:
Overall Officials: I-Te Lee, MD,PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Division of Endocrinology and Metabolism in Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Not to share individual participant data